CLINICAL TRIAL: NCT04012294
Title: Effects of Allopurinol on Inflammatory Markers and Morphostructural Changes Evidenced by Musculoskeletal Ultrasound in Individuals With Asymptomatic Hyperuricemia. A Proof of Concept
Brief Title: Effects of Allopurinol on Inflammation and Ultrasonographic Changes in People With Elevated Uric Acid But no Symptoms
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Collaborators: Instituto Nacional de Rehabilitacion (Other Government)
Responsible Party: Principal Investigator, Luis M Amezcua-Guerra, Head of Immunology Department, Principal Investigator, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CardiologiaIC
Record Dates: First submitted 2019-07-03; First posted 2019-07-09 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Musculoskeletal Degeneration; Inflammation; Hyperuricemia
Keywords: allopurinol; ultrasound; morphostructural changes
MeSH Terms: conditions — Inflammation; Hyperuricemia | interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- allopurinol (Experimental): 150 mg daily for a month then 300 mg daily for the rest of the study (5 months)
  Interventions: Drug: Allopurinol Pill

INTERVENTIONS:
Drug: Allopurinol Pill — Individuals who meet the inclusion criteria and also have morphostructural changes suggestive of MSU crystal deposits in their MSUS will start treatment with allopurinol at a dosage of 150 mg to be taken daily, orally for a month and then to be increased to 300 mg. The rest of the individuals' medication is not to be altered. If a participant presents hypersensitivity to allopurinol, they are to stop the medication and will be excluded from the investigation.
  Three months after starting treatment, the participants will have a physical exam, confirm the continuation of the treatment (adjust dosage if needed) and take a blood sample for laboratory tests. Six months after treatment is started, the participants will be reevaluated by MSUS and have another blood sample taken, Once the study is finished, continuing or ending treatment with allopurinol will be decided by the medical judgment of the physician of each participant.
  Other Names: Zyloprim

SUMMARY:
Hyperuricemia is a metabolic alteration defined as the presence of serum urate levels higher than 7 mg/dL. This has proven to be the maximum limit of solubility of urate in serum, any higher concentration leads to precipitation and eventually to the formation of monosodium urate (MSU) crystals. The accumulation of said crystals can manifest as gouty arthritis, uric acid nephropathy, urolithiasis or chronic tophaceous gout.

A strong relation between hyperuricemia and other chronic degenerative diseases, including diabetes mellitus, systemic arterial hypertension, obesity and metabolic syndrome, has been consistently proven.

Hypouricemic pharmacological agents have shown a decrease in cardiovascular complications and death in patients with gout.

A series of studies conducted on individuals with asymptomatic hyperuricemia using musculoskeletal ultrasound (MSUS) have shown the presence of morphostructural changes suggestive of MSU crystal deposits, combined with an elevation in a series of inflammation markers to a degree similar to those found in patients with chronic gout.

Even though, there is evidence of morphostructural damage in individuals with asymptomatic hyperuricemia, there are no clinical, laboratorial or imaging parameters that indicate when hypouricemic treatment should be started.

This clinical trial is proposed as a proof of concept which is looking to evaluate if treatment with allopurinol induces changes in levels of inflammatory markers in individuals with asymptomatic hyperuricemia and morphostructural changes suggestive of MSU crystal deposits. this proof of concept is not looking to measure the efficiency, effectiveness or security of the treatment.

Our Hypothesis is that Individuals with asymptomatic hyperuricemia and morphostructural changes evidenced by MSUS (double contour sing, tophi, aggregates) will show a decent in inflammatory markers and their morphostructural changes will diminish or revert after treatment with allopurinol.

DETAILED DESCRIPTION:
Gout is the most prevalent inflammatory rheumatological disease among young men, affecting about 4% of the general population. Caused by the deposit of monosodium urate (MSU) crystals which form because of high urate concentrations in serum. Currently, there is no universal definition for hyperuricemia but The Gout, Hyperuricemia, and Crystal-Associated Disease Network (G-CAN) define hyperuricemia as a blood urate concentration above the saturation threshold which is usually understood to be urate levels over 7 mg/dL. For this study, the term urate will be used as the final circulating product of the enzyme xanthine oxidase in the purine metabolism which favors the precipitation and formation of MSU crystals. Even tough, hyperuricemia is often asymptomatic, the clinical presentation can be that of gouty arthritis, uric acid nephropathy, urolithiasis and/or chronic tophaceous gout.

The relevance of asymptomatic hyperuricemia lays in the relation to other chronic degenerative diseases, including atherosclerotic disease, systemic arterial hypertension, coronary artery disease and chronic kidney disease.

A logistic regression analysis made by Zhu et al, looking specifically at the demographics of gout and asymptomatic hyperuricemia based on the data from The National Health and Nutrition Examination Survey (NHANES) showed a general hyperuricemia prevalence of 13.2%, which corresponds to about 26.6 million individuals. Additionally, it was observed that hyperuricemia increases with age, it being more common in individuals over 65 years, prevalence of 31%, corresponding to approximately 10.7 million American adults. Other epidemiological studies have evidenced the relationship between asymptomatic hyperuricemia y different comorbidities for example atherosclerotic disease, systemic arterial hypertension, coronary artery disease and metabolic syndrome. Those studies suggest that elevated urate levels are an independent cardiovascular risk factor. Their findings also suggest that lowering serum urate levels is associated with a descend in the risk of cardiovascular complications. In spite of this, there is currently no indication for hypouricemic pharmacological treatment for individuals with hyperuricemia that don´t have a diagnosis of gout, urolithiasis, uric acid nephropathy or as prophylaxis for tumoral lysis syndrome. The I-Lan Longitudinal Aging Study (ILAS), a cohort study from Taiwan, showed a higher cardiovascular risk in individuals without diabetes or previous cardiovascular disease but with serum urate levels above 6.1 mg/dL. Lastly, our group has shown that the presence of hyperuricemia at admission in the emergency room doubles the short-term risk of death (30 days) in patients with coronary heart disease.

Hyperuricemia increases the risk of atherosclerosis by up to 60%. It is believed that the cause for this lay in the activation of the inflammasome´s cryopyrin (NLRP3) protein complex by the MSU crystals . This promotes the release of pro-inflammatory cytokines and chemokines, particularly the mature forms of interleukin (IL)-1β and IL-18. In addition, the phagocytosis of MSU crystals executed by neutrophils and macrophages, induces production of reactive oxygen and nitrogen species all of which lead to oxidative stress and consequently to endothelial dysfunction. When kept chronically, it is probable that these mechanisms result in atherosclerosis. Solid evidence has shown that pharmacological treatment aimed at reducing urate levels is beneficial in patients with gout since it lowers the occurrence of adverse cardiovascular events and all-cause mortality. There is still a group of individuals with chronically elevated urate levels without clinical manifestations for which pharmacological treatment remains a topic of debate and controversy. Even though, some of these individuals could benefit from hypouricemic pharmacological therapy, there is currently no criteria for determining when it should be started. The first line of treatment are xanthine oxidase inhibitors like allopurinol and febuxostat. Both lower serum urate in comparable concentrations but a study done comparing the two agents showed that allopurinol induces a more significant global survival rate than febuxostat therefore treatment with allopurinol is preferred.

Musculoskeletal ultrasound (MSUS) has proven to be an excellent, noninvasive, diagnostic tool for different articular and rheumatological diseases. Its value lays in the evaluation of tendons, ligaments, joints and periarticular soft tissue. MSUS is useful in early stages of a disease, when no symptoms are present, and also at the chronic stages with established morphostructural damage. It has proven to be sensible to change, so it can be used to follow up on morphostructural changes during the course of treatment. Additionally, having color doppler and power doppler (PD) technology allows for the visualization of the degree of vascularization and angiogenesis in the affected tissue. These are the reasons MSUS is considered an innocuous imaging method which works without radiation, that is less costly and more accessible than most other imaging technologies. A series of studies show the relevance of MSUS for the detection of morphostructural changes suggestive of MSU deposits characteristically found in gout. The ultrasonographic signs related to said deposits are hyperechoic enhancement of the superficial margin of the hyaline cartilage, better known as the double contour sign, widening of the joint cavity, aggregates, tophi, and erosions. Wright et al compared MSUS´ and conventional radiography's capacity to detect erosions secondary to gout on the first metatarsophalangeal joint of 78 patients. MSUS proved to be superior in that study.

In previous studies, our group has observed the presence of morphostructural changes suggestive of MSU deposits in individuals with asymptomatic hyperuricemia using MSUS. The change observed in the joints was similar to that of patients with a gout diagnosis. The main findings were hyperechoic enhancement of the superficial margin of the hyaline cartilage (double contour sign) on the femoral cartilage and first metatarsophalangeal joint, intraarticular tophi, as well as patellar and Achilles enthesopathy. These results have since been replicated even in animal models, supporting that asymptomatic hyperuricemia induces morphostructural changes in different tissues (hyaline cartilage, entheses, tendons and subchondral bone) before leading to an acute gout attack or an episode of urolithiasis.

Recently, our group investigated a possible association between morphostructural changes suggestive of MSU deposits and the elevation of inflammation markers in individuals with asymptomatic hyperuricemia. For this purpose, three groups were studied: the first made up of individuals with asymptomatic hyperuricemia, the second formed by patients with chronic gout, and the third comprised of normouricemic individuals as a control group. All participants got an MSUS of the knee, ankle and first metatarsophalangeal joint in search for morphostructural changes suggestive of MSU deposits. The serum concentrations of IL-1β, IL-2, IL-4, IL-5, IL-6, IL- 10, IL-12, IL-13, interferon -γ(INF) and tumoral necrosis factor (TNF) were measured in all the participants. The levels of the following chemokines IL-8 also known as C-X-C Motif chemokine ligand 8 (CXCL8), monocyte chemoattractant protein 1 (MCP-1) also known as C-C Motif Chemokine Ligand 2 (CCL2) and epithelial-derived neutrophil-activating peptide 78 (ENA-78) also known as C-X-C Motif chemokine ligand 5 (CXCL5), and microRNA(miR) miR-146a, miR-155 y miR-223 were also quantified.

In this study, the investigators found that individuals with asymptomatic hyperuricemia present similar levels of cytokines and chemokines as those observed in patients with gout; more notably the serum concentration of IL-6, IL-8 and miR-155 were significantly higher in both groups when compared to the normouricemic controls. Also, a significant relation between presence of MSU crystals (independent of urate acid levels) and higher levels of IL-6, IL-8 and miR-155 was found. This is the first study to suggest that the presence of MSU deposits (detected by MSUS) are a marker of inflammatory activity independent of the existence or lack of previous gouty arthritis episodes.

The elevated levels of inflammatory cytokines, chemokines and microRNA in individuals with asymptomatic hyperuricemia makes questioning the need for pharmacological treatment in this group even more relevant.

The more knowledge is gained on the beginning and progression of atherosclerotic heart disease, the more evident it becomes that local and systemic inflammatory processes are associated.

Chronic, systemic inflammation can be evidenced by different premature immunosenescence phenomena, among them the loss of expression of the co-signalizing Cluster of Differentiation 28(CD 28) molecule from T CD4 + lymphocytes is of particular interest. The percentage of Cluster of Differentiation 4 that lack the expression of Cluster of Differentiation 28 (CD4+ CD28null) is a relievable marker that is sensible to change of chronic inflammation and atherosclerotic damage.

As a matter of fact, the presence of activated systemic inflammatory pathways could be the etiopathogenic bond that unites a persistent elevation of urate serum concentration with the development of accelerated atherosclerosis and adverse cardiovascular events including coronary artery disease. By this logic, individuals with asymptomatic hyperuricemia with evidence of MSU articular deposits are the ones that could benefit from hypouricemic treatment since this would lower local and systemic inflammation.

A score which can be used to predict the risk of myocardial infarction or stroke (QRISK3). The variables it uses are age, gender, ethnicity, tobacco consumption, previous diagnostic of diabetes, chronic kidney disease, rheumatoid arthritis, systemic lupus erythematosus or severe psychiatric disease; family history of angina or myocardial infarction before 60 years of age, use of drugs for erectile disfunction, antihypertensives, atypical antipsychotics or regular use of steroids, and body mass index. Its algorithm provides four results: 10-year risk given as a percentage, the result a healthy person of the same age, gender and ethnicity would get, relative risk, and the age at which a healthy individual would have the same risk as the patient.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with two urate determinations >7 mg/dL in the last year and no clinical sign, past or present, suggestive of joint inflammation (acute gout attack), urolithiasis or uric acid nephropathy
* Over 18 years of age
* Residents of Mexico City or its metropolitan area
* Individuals with a signed informed consent form for the participation in the clinical trial

Exclusion Criteria:

* Individuals with joint inflammation suggestive of gout during the clinical evaluation
* Patients without elemental ultrasonographic lesions (double contour sign, aggregates, tophi) on the first metatarsophalangeal joint, knee, ankle or the tendons of the quadriceps, patella, and calcaneus when evaluated by MSUS
* Patients taking thiazides
* Patients with history of stroke or coronary artery disease in the last year
* Patients with osteoarthritis be it by clinical presentation or imaging
* Pregnant women
* Neoplasms
* Known Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) , Human immunodeficiency Virus (HIV) infection, or any other know active infections
* Autoimmune or autoinflammatory disease
* Allopurinol hypersensitivity or allergy
* Deteriorated kidney function (Glomerular Filtration Rate (GFR) <50 mL/min/1.73m^2)
* Patients taking azathioprine
* Functional New York Heart Association (NYHA) score of II or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-08-30 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
inflammatory markers | 6 months
  To measure changes in proinflammatory cytokines (Interleukin 1ß (IL-1ß))
inflammatory markers | 6 months
  To measure changes in proinflammatory cytokines (Tumor Necrosis Factor)
inflammatory markers | 6 months
  To measure changes in proinflammatory cytokines (Interleukin 6 (IL-6))
inflammatory markers | 6 months
  To measure changes in proinflammatory cytokines (Interferon-γ)
inflammatory markers | 6 months
  To measure changes in proinflammatory cytokines (Interleukin 18 (IL-18))
inflammatory markers | 6 months
  To measure changes in proinflammatory cytokines (Interleukin 17 (IL-17))
inflammatory markers | 6 months
  To measure changes in chemokines (Interleukin 8 (IL-8))
inflammatory markers | 6 months
  To measure changes in chemokines (monocyte chemoattractant protein 1 (MCP-1))
inflammatory markers | 6 months
  To measure changes in microRNAs (miR) (miR-155)
inflammatory markers | 6 months
  To measure changes in the percentage of Cluster of Differentiation 4 cells that lack the expression of Cluster of Differentiation 28 (CD4+CD28null)

SECONDARY OUTCOMES:
musculoskeletal ultrasound | 6 months
  Presence of the ultrasonographic elemental lesions caused by monosodium urate crystals: (Double contour sign is a hyperechoic abnormal band over the superficial margin of articular hyaline cartilage, independent from insonation angle which can be regular or irregular, continuous or intermittent and that distinguishes itself from the cartilage interphase sign)
musculoskeletal ultrasound | 6 months
  Presence of the ultrasonographic elemental lesions caused by monosodium urate crystals: (Tophi are described, independent of location, as an heterogenous, circumscript aggregate, hyper- and/or hypoechoic, which can be surrounded by a small anechoic halo and can have a posterior acoustic shadow)
musculoskeletal ultrasound | 6 months
  Presence of the ultrasonographic elemental lesions caused by monosodium urate crystals: (Aggregates are described, independent of location, as heterogenous hyperechoic foci which maintain a high degree of reflectivity even when gain is reduced to the minimum or when the insonation angle is changed, also they can sometimes create a posterior acoustic shadow)
musculoskeletal ultrasound | 6 months
  Presence of the ultrasonographic elemental lesions caused by monosodium urate crystals: (Erosions are described as a discontinuation of the bone surface, seen in two perpendicular planes)

CONTACTS AND LOCATIONS:
Overall Officials: Luis M Amezcua-Guerra, MD, Principal Investigator — Instituto Nacional de Cardiologia Ignacio Chavez
Locations (2):
- Mexico (2):
  - Instituto Nacional de Cardiología, Mexico City
  - National Institute of Cardiology Mexico, Mexico City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang W, Doherty M, Bardin T, Pascual E, Barskova V, Conaghan P, Gerster J, Jacobs J, Leeb B, Liote F, McCarthy G, Netter P, Nuki G, Perez-Ruiz F, Pignone A, Pimentao J, Punzi L, Roddy E, Uhlig T, Zimmermann-Gorska I; EULAR Standing Committee for International Clinical Studies Including Therapeutics. EULAR evidence based recommendations for gout. Part II: Management. Report of a task force of the EULAR Standing Committee for International Clinical Studies Including Therapeutics (ESCISIT). Ann Rheum Dis. 2006 Oct;65(10):1312-24. doi: 10.1136/ard.2006.055269. Epub 2006 May 17. PMID 16707532
- [Background] Bursill D, Taylor WJ, Terkeltaub R, Kuwabara M, Merriman TR, Grainger R, Pineda C, Louthrenoo W, Edwards NL, Andres M, Vargas-Santos AB, Roddy E, Pascart T, Lin CT, Perez-Ruiz F, Tedeschi SK, Kim SC, Harrold LR, McCarthy G, Kumar N, Chapman PT, Tausche AK, Vazquez-Mellado J, Gutierrez M, da Rocha Castelar-Pinheiro G, Richette P, Pascual E, Fisher MC, Burgos-Vargas R, Robinson PC, Singh JA, Jansen TL, Saag KG, Slot O, Uhlig T, Solomon DH, Keenan RT, Scire CA, Biernat-Kaluza E, Dehlin M, Nuki G, Schlesinger N, Janssen M, Stamp LK, Sivera F, Reginato AM, Jacobsson L, Liote F, Ea HK, Rosenthal A, Bardin T, Choi HK, Hershfield MS, Czegley C, Choi SJ, Dalbeth N. Gout, Hyperuricemia, and Crystal-Associated Disease Network Consensus Statement Regarding Labels and Definitions for Disease Elements in Gout. Arthritis Care Res (Hoboken). 2019 Mar;71(3):427-434. doi: 10.1002/acr.23607. PMID 29799677
- [Background] Paul BJ, Anoopkumar K, Krishnan V. Asymptomatic hyperuricemia: is it time to intervene? Clin Rheumatol. 2017 Dec;36(12):2637-2644. doi: 10.1007/s10067-017-3851-y. Epub 2017 Oct 4. PMID 28980141
- [Background] Campion EW, Glynn RJ, DeLabry LO. Asymptomatic hyperuricemia. Risks and consequences in the Normative Aging Study. Am J Med. 1987 Mar;82(3):421-6. doi: 10.1016/0002-9343(87)90441-4. PMID 3826098
- [Background] Zhu Y, Pandya BJ, Choi HK. Prevalence of gout and hyperuricemia in the US general population: the National Health and Nutrition Examination Survey 2007-2008. Arthritis Rheum. 2011 Oct;63(10):3136-41. doi: 10.1002/art.30520. PMID 21800283
- [Background] Feig DI, Kang DH, Johnson RJ. Uric acid and cardiovascular risk. N Engl J Med. 2008 Oct 23;359(17):1811-21. doi: 10.1056/NEJMra0800885. No abstract available. PMID 18946066
- [Background] Wu MY, Li CJ, Hou MF, Chu PY. New Insights into the Role of Inflammation in the Pathogenesis of Atherosclerosis. Int J Mol Sci. 2017 Sep 22;18(10):2034. doi: 10.3390/ijms18102034. PMID 28937652
- [Background] Edwards NL. The role of hyperuricemia and gout in kidney and cardiovascular disease. Cleve Clin J Med. 2008 Jul;75 Suppl 5:S13-6. doi: 10.3949/ccjm.75.suppl_5.s13. PMID 18822470
- [Background] Chang CC, Wu CH, Liu LK, Chou RH, Kuo CS, Huang PH, Chen LK, Lin SJ. Association between serum uric acid and cardiovascular risk in nonhypertensive and nondiabetic individuals: The Taiwan I-Lan Longitudinal Aging Study. Sci Rep. 2018 Mar 27;8(1):5234. doi: 10.1038/s41598-018-22997-0. PMID 29588485
- [Background] Mora-Ramirez M, Estevez-Garcia IO, Irigoyen-Camacho ME, Bojalil R, Gonzalez-Pacheco H, Amezcua-Guerra LM. Hyperuricemia on Admission Predicts Short-Term Mortality due to Myocardial Infarction in a Population with High Prevalence of Cardiovascular Risk Factors. Rev Invest Clin. 2017 Sep-Oct;69(5):247-253. doi: 10.24875/ric.17002167. PMID 29077696
- [Background] Kushiyama A, Nakatsu Y, Matsunaga Y, Yamamotoya T, Mori K, Ueda K, Inoue Y, Sakoda H, Fujishiro M, Ono H, Asano T. Role of Uric Acid Metabolism-Related Inflammation in the Pathogenesis of Metabolic Syndrome Components Such as Atherosclerosis and Nonalcoholic Steatohepatitis. Mediators Inflamm. 2016;2016:8603164. doi: 10.1155/2016/8603164. Epub 2016 Dec 14. PMID 28070145
- [Background] Zamudio-Cuevas Y, Martinez-Flores K, Fernandez-Torres J, Loissell-Baltazar YA, Medina-Luna D, Lopez-Macay A, Camacho-Galindo J, Hernandez-Diaz C, Santamaria-Olmedo MG, Lopez-Villegas EO, Oliviero F, Scanu A, Cerna-Cortes JF, Gutierrez M, Pineda C, Lopez-Reyes A. Monosodium urate crystals induce oxidative stress in human synoviocytes. Arthritis Res Ther. 2016 May 21;18(1):117. doi: 10.1186/s13075-016-1012-3. PMID 27209322
- [Background] Rada B. Neutrophil Extracellular Traps and Microcrystals. J Immunol Res. 2017;2017:2896380. doi: 10.1155/2017/2896380. Epub 2017 Mar 7. PMID 28373994
- [Background] Stamp L, Dalbeth N. Urate-lowering therapy for asymptomatic hyperuricaemia: A need for caution. Semin Arthritis Rheum. 2017 Feb;46(4):457-464. doi: 10.1016/j.semarthrit.2016.07.015. Epub 2016 Jul 28. PMID 27591828
- [Background] Chales G. How should we manage asymptomatic hyperuricemia? Joint Bone Spine. 2019 Jul;86(4):437-443. doi: 10.1016/j.jbspin.2018.10.004. Epub 2018 Oct 11. PMID 30316974
- [Background] White WB, Saag KG, Becker MA, Borer JS, Gorelick PB, Whelton A, Hunt B, Castillo M, Gunawardhana L; CARES Investigators. Cardiovascular Safety of Febuxostat or Allopurinol in Patients with Gout. N Engl J Med. 2018 Mar 29;378(13):1200-1210. doi: 10.1056/NEJMoa1710895. Epub 2018 Mar 12. PMID 29527974
- [Background] Filippucci E, Scire CA, Delle Sedie A, Iagnocco A, Riente L, Meenagh G, Gutierrez M, Bombardieri S, Valesini G, Montecucco C, Grassi W. Ultrasound imaging for the rheumatologist. XXV. Sonographic assessment of the knee in patients with gout and calcium pyrophosphate deposition disease. Clin Exp Rheumatol. 2010 Jan-Feb;28(1):2-5. PMID 20346230
- [Background] Ventura-Rios L, Sanchez-Bringas G, Pineda C, Hernandez-Diaz C, Reginato A, Alva M, Audisio M, Bertoli A, Cazenave T, Gutierrez M, Mora C, Py G, Sedano O, Solano C, de Miguel E. Tendon involvement in patients with gout: an ultrasound study of prevalence. Clin Rheumatol. 2016 Aug;35(8):2039-2044. doi: 10.1007/s10067-016-3309-7. Epub 2016 May 28. PMID 27236513
- [Background] Pineda C, Amezcua-Guerra LM, Solano C, Rodriguez-Henriquez P, Hernandez-Diaz C, Vargas A, Hofmann F, Gutierrez M. Joint and tendon subclinical involvement suggestive of gouty arthritis in asymptomatic hyperuricemia: an ultrasound controlled study. Arthritis Res Ther. 2011 Jan 17;13(1):R4. doi: 10.1186/ar3223. PMID 21241475
- [Background] Wright SA, Filippucci E, McVeigh C, Grey A, McCarron M, Grassi W, Wright GD, Taggart AJ. High-resolution ultrasonography of the first metatarsal phalangeal joint in gout: a controlled study. Ann Rheum Dis. 2007 Jul;66(7):859-64. doi: 10.1136/ard.2006.062802. Epub 2006 Dec 21. PMID 17185326
- [Background] Viggiano D, Gigliotti G, Vallone G, Giammarino A, Nigro M, Capasso G. Urate-Lowering Agents in Asymptomatic Hyperuricemia: Role of Urine Sediment Analysis and Musculoskeletal Ultrasound. Kidney Blood Press Res. 2018;43(2):606-615. doi: 10.1159/000489145. Epub 2018 Apr 19. PMID 29689561
- [Background] Pineda C, Fuentes-Gomez AJ, Hernandez-Diaz C, Zamudio-Cuevas Y, Fernandez-Torres J, Lopez-Macay A, Alba-Sanchez I, Camacho-Galindo J, Ventura L, Gomez-Quiroz LE, Gutierrez-Ruiz MC, Garcia-Vazquez F, Reginato AM, Gutierrez M, Lopez-Reyes A. Animal model of acute gout reproduces the inflammatory and ultrasonographic joint changes of human gout. Arthritis Res Ther. 2015 Feb 26;17(1):37. doi: 10.1186/s13075-015-0550-4. PMID 25889158
- [Background] Puig JG, Beltran LM, Mejia-Chew C, Tevar D, Torres RJ. Ultrasonography in the diagnosis of asymptomatic hyperuricemia and gout. Nucleosides Nucleotides Nucleic Acids. 2016 Dec;35(10-12):517-523. doi: 10.1080/15257770.2015.1124999. PMID 27906639
- [Background] Estevez-Garcia IO, Gallegos-Nava S, Vera-Perez E, Silveira LH, Ventura-Rios L, Vancini G, Hernandez-Diaz C, Sanchez-Munoz F, Ballinas-Verdugo MA, Gutierrez M, Pineda C, Rodriguez-Henriquez P, Castillo-Martinez D, Amezcua-Guerra LM. Levels of Cytokines and MicroRNAs in Individuals With Asymptomatic Hyperuricemia and Ultrasonographic Findings of Gout: A Bench-to-Bedside Approach. Arthritis Care Res (Hoboken). 2018 Dec;70(12):1814-1821. doi: 10.1002/acr.23549. Epub 2018 Nov 2. PMID 29457379
- [Background] Crea F, Libby P. Acute Coronary Syndromes: The Way Forward From Mechanisms to Precision Treatment. Circulation. 2017 Sep 19;136(12):1155-1166. doi: 10.1161/CIRCULATIONAHA.117.029870. PMID 28923905
- [Background] Dumitriu IE. The life (and death) of CD4+ CD28(null) T cells in inflammatory diseases. Immunology. 2015 Oct;146(2):185-93. doi: 10.1111/imm.12506. Epub 2015 Sep 7. PMID 26190355
- [Background] Gutierrez M, Schmidt WA, Thiele RG, Keen HI, Kaeley GS, Naredo E, Iagnocco A, Bruyn GA, Balint PV, Filippucci E, Mandl P, Kane D, Pineda C, Delle Sedie A, Hammer HB, Christensen R, D'Agostino MA, Terslev L; OMERACT Ultrasound Gout Task Force group. International Consensus for ultrasound lesions in gout: results of Delphi process and web-reliability exercise. Rheumatology (Oxford). 2015 Oct;54(10):1797-805. doi: 10.1093/rheumatology/kev112. Epub 2015 May 13. PMID 25972391
- [Background] Wakefield RJ, Gibbon WW, Conaghan PG, O'Connor P, McGonagle D, Pease C, Green MJ, Veale DJ, Isaacs JD, Emery P. The value of sonography in the detection of bone erosions in patients with rheumatoid arthritis: a comparison with conventional radiography. Arthritis Rheum. 2000 Dec;43(12):2762-70. doi: 10.1002/1529-0131(200012)43:123.0.CO;2-#. PMID 11145034
- [Background] D'Agostino MA, Terslev L, Aegerter P, Backhaus M, Balint P, Bruyn GA, Filippucci E, Grassi W, Iagnocco A, Jousse-Joulin S, Kane D, Naredo E, Schmidt W, Szkudlarek M, Conaghan PG, Wakefield RJ. Scoring ultrasound synovitis in rheumatoid arthritis: a EULAR-OMERACT ultrasound taskforce-Part 1: definition and development of a standardised, consensus-based scoring system. RMD Open. 2017 Jul 11;3(1):e000428. doi: 10.1136/rmdopen-2016-000428. eCollection 2017. PMID 28948983
- [Background] Xiang M, Zeng Y, Yang R, Xu H, Chen Z, Zhong J, Xie H, Xu Y, Zeng X. U6 is not a suitable endogenous control for the quantification of circulating microRNAs. Biochem Biophys Res Commun. 2014 Nov 7;454(1):210-4. doi: 10.1016/j.bbrc.2014.10.064. Epub 2014 Oct 18. PMID 25450382
- [Background] Shen J, Todd NW, Zhang H, Yu L, Lingxiao X, Mei Y, Guarnera M, Liao J, Chou A, Lu CL, Jiang Z, Fang H, Katz RL, Jiang F. Plasma microRNAs as potential biomarkers for non-small-cell lung cancer. Lab Invest. 2011 Apr;91(4):579-87. doi: 10.1038/labinvest.2010.194. Epub 2010 Nov 29. PMID 21116241
- [Background] Hippisley-Cox J, Coupland C, Brindle P. Development and validation of QRISK3 risk prediction algorithms to estimate future risk of cardiovascular disease: prospective cohort study. BMJ. 2017 May 23;357:j2099. doi: 10.1136/bmj.j2099. PMID 28536104
- [Derived] Amezcua-Guerra LM, Espinosa-Bautista F, Hopf-Estandia K, Valdivieso-Ruiz M, Coronel D, Robledo S, Ramos-Rosillo V, Del Rocio Martinez-Alvarado M, Patlan M, Paez A, Silveira LH, Tavera-Alonso C, Masso F, Soto-Fajardo C, Pineda C. Senescent CD4+CD28null cells are increased in chronic hyperuricemia, show aberrant effector phenotypes, and are reversed after allopurinol therapy: a proof-of-concept pilot study. Clin Rheumatol. 2023 Aug;42(8):2181-2186. doi: 10.1007/s10067-023-06595-8. Epub 2023 Apr 18. PMID 37072512